CLINICAL TRIAL: NCT00433121
Title: Discontinuation of Antipsychotics and Antidepressants Among Patients With Dementia and BPSD Living in Nursing Homes - an Open Study.
Brief Title: Discontinuation of Antipsychotics and Antidepressants Among Patients With BPSD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Demensforbundet, Norway (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101
Record Dates: First submitted 2007-02-01; First posted 2007-02-09 (Estimated); Last update posted 2007-08-24 (Estimated); Status verified 2007-08

CONDITIONS: Dementia
Keywords: Antidepressive Agents; Neuroleptica; Dementia; Discontinuation study; Behavioural- and Psychological Symptoms in Dementia
MeSH Terms: conditions — Dementia | interventions — Risperidone; Olanzapine; Escitalopram; Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Discontinuation of neuroleptic or anti depressants
  Interventions: Drug: Risperidone; Drug: Olanzapine; Drug: Haloperidole; Drug: Quetiapin; Drug: Escitalopram; Drug: Citalopram; Drug: Sertralin

INTERVENTIONS:
Drug: Risperidone
Drug: Olanzapine
Drug: Haloperidole
Drug: Quetiapin
Drug: Escitalopram
Drug: Citalopram
Drug: Sertralin

SUMMARY:
The aim of this study is to discontinue antipsychotics and antidepressants, and to study its effect on Behavioural- and Psychological Symptoms in Dementia (BPSD).

DETAILED DESCRIPTION:
Patients with dementia have cognitive deficits, but also hallucinations, delusions, agitation, aggression and apathy. These symptoms are called Behavioural- and Psychological Symptoms in Dementia (BPSD), and are difficult to treat. Antipsychotic and antidepressant medication is in use, despite its lack of clinical evidence.

We will discontinue antipsychotics in one group of 12 patients and antidepressants in one group of 12 patients. Patients should have dementia of Alzheimer- or vascular origin. They should live in Nursing Homes and have no other psychiatric disease for which they receive psychotropic drug. They will be registered with 7 different questionnaires at baseline and after 3, 6, 12 and 24 weeks. The study period is 24 weeks. The questionnaires are filled in by the patients and the nurses at the nursing homes.

This is an open labelled study with no control group. Based on the results of this study, we will design a RCT study with placebo-controlled group.

ELIGIBILITY:
Inclusion Criteria:

* Vascular- or Alzheimer Dementia
* Nursing Homes resident for 3 months or more
* Given antipsychotics or antidepressants for 3 months or more
* Clinical Dementia rating 1, 2 or 3

Exclusion Criteria:

* Dementia of other origin
* Psychiatric disease
* Life expectancy less than 3 months
* Acute infection last 10 days
* Unstable Diabetes Mellitus
* Terminal disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Changes in Neuropsychiatric Inventory | 24 weeks
Changes in weight | 24 weeks
Changes in Cornell's Depression Scale | 24 weeks
Changes in UPDRS subscale | 24 weeks
Changes in "Quality of Live - Alzheimer Disease" | 24 weeks

SECONDARY OUTCOMES:
Changes in Severe Impairment Battery | 24 weeks
Changes in Lawton's PADL | 24 weeks
Oxazepam given p.n. | 24 weeks
Drop outs | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Knut Engedal, Ph D, Study Chair — The Norwegian Centre for Dementia Research (NCDR), Norway
Locations (1):
- Sykehuset Innlandet HF - Sanderud, Ottestad, Oppland, Norway